CLINICAL TRIAL: NCT04511611
Title: Randomized, Non-blinded, Two-way Crossover Study to Assess Bioequivalence Between a Rivaroxaban 10 mg Orally Disintegrating Tablet Administered With Water or Without Water and a Rivaroxaban 10 mg Film-coated Tablet in Japanese Healthy Male Adult Subjects
Brief Title: Study to Compare the Effect of the Formulations (Orally Disintegrating Tablet and Film-coated Tablet) on Bioequivalence of Drug Rivaroxaban (Xarelto) at Dose of 10 mg in Japanese Healthy Male Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20087
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test A: 10 mg ODT with water, then 10 mg film-coated tablet (Experimental): Participants received one single dose of 10 mg rivaroxaban orally disintegrating tablet (ODT) with water in the fasted state. After a washing period of 5 days, participants received one single oral dose of 10 mg rivaroxaban film-coated tablet in the fasted state
  Interventions: Drug: Rivaroxaban (BAY 59-7939, Xarelto) in ODT form; Drug: Rivaroxaban (BAY 59-7939, Xarelto) in film-coated form
- Test A: 10 mg film-coated tablet, then 10 mg ODT with water (Experimental): Participants received one single dose of 10 mg rivaroxaban film-coated tablet in the fasted state. After a washing period of 5 days, participants received one single oral dose of 10 mg rivaroxaban orally disintegrating tablet (ODT) with water in the fasted state
  Interventions: Drug: Rivaroxaban (BAY 59-7939, Xarelto) in ODT form; Drug: Rivaroxaban (BAY 59-7939, Xarelto) in film-coated form
- Test B: 10 mg ODT without water, then 10 film-coated tablet (Experimental): Participants received one single dose of 10 mg rivaroxaban orally disintegrating tablet (ODT) without water in the fasted state. After a washing period of 5 days, participants received one single oral dose of 10 mg rivaroxaban film-coated tablet in the fasted state
  Interventions: Drug: Rivaroxaban (BAY 59-7939, Xarelto) in ODT form; Drug: Rivaroxaban (BAY 59-7939, Xarelto) in film-coated form
- Test B: 10 mg film-coated tablet, then 10 mg ODT without water (Experimental): Participants received one single dose of 10 mg rivaroxaban film-coated tablet in the fasted state. After a washing period of 5 days, participants received one single oral dose of 10 mg rivaroxaban orally disintegrating tablet (ODT) without water in the fasted state
  Interventions: Drug: Rivaroxaban (BAY 59-7939, Xarelto) in ODT form; Drug: Rivaroxaban (BAY 59-7939, Xarelto) in film-coated form

INTERVENTIONS:
Drug: Rivaroxaban (BAY 59-7939, Xarelto) in ODT form — 10 mg as 1 x 10 mg orally disintegrating tablet (ODT)
Drug: Rivaroxaban (BAY 59-7939, Xarelto) in film-coated form — 10 mg as 1 x 10 mg film-coated tablet

SUMMARY:
Researchers in this study wanted to compare the effect of the formulation (orally disintegrating tablet and film-coated tablet) on the bioequivalence of drug Rivaroxaban (brand name: Xarelto) at dose of 10 mg in Japanese healthy male subjects aged 20 to 40 years. Rivaroxaban is an approved drug to be used for the prevention of events/diseases caused by blood clots. Currently, there are two formulations of Rivaroxaban available on the market in Japan and they are film-coated tablets and fine granules. To further improve patients' convenience, a new formulation, orally disintegrating tablet (ODT, a drug dosage form designed to be dissolved on the tongue rather than swallowed whole) is under development. The goal of this study was to compare the effect of this new formulation with film-coated tablets when taken with or without water.

Participants in this study received one oral dose of rivaroxaban 10 mg ODT either with or without water and one oral dose of rivaroxaban 10 mg film-tablet. There were at least 5 days between the two doses. Observation for each participant lasted about 6 weeks in total. Blood samples were collected from the participants to measure the blood level of the study drug.

ELIGIBILITY:
Inclusion Criteria:

- Japanese healthy male subjects, aged 20 to 40 years (inclusive), with body mass index 17.6 to 26.4 kg/m²

Exclusion Criteria:

* Subject with incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study drugs will not be normal
* Subject with known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Subject with known coagulation disorders (e.g. von Willebrand disease, hemophilia)
* Subject with febrile illness within 1 week before the first study drug administration
* Subject with suspicion of drug or alcohol abuse
* Subject with intake of foods or beverages containing grapefruit, pomelo, Seville orange, and tangelo within 1 week before the first study drug administration
* Subject with therapies (e.g. physiotherapy, acupuncture, etc.) within 1 month before starting study treatment
* Subject with clinically relevant findings in the electrocardiogram (ECG) such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over 120 msec or of the corrected QT (QTc) interval over 450 msec
* Subject with systolic blood pressure below 90 or above 130 mmHg
* Subject with diastolic blood pressure below 45 or above 85 mmHg
* Subject with clinically relevant deviations of the screened laboratory parameters from reference ranges

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Cmax for plasma rivaroxaban concentration | Up to 48 hours after study medication
  Maximum observed concentration
AUC(0-tlast) for plasma rivaroxaban concentration | Up to 48 hours after study medication
  Area under the concentration versus time curve from time 0 to the last data point > lower limit of quantitation

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events | Up to 30 days after study medication

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Sumida Hospital, Sumida-ku, Tokyo
  - Fukuoka Mirai Hospital, Fukuoka
  - Medical Co. LTA Nishikumamoto hospital, Kumamoto

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/